CLINICAL TRIAL: NCT03023462
Title: Efficacy of the Anterior Quadratus Lumborum Block Versus the Transversus Abdominis Plane Block for Elective Laparoscopic Inguinal Hernia Repair: A Randomized Controlled Trial
Brief Title: Efficacy of an Anterior Quadratus Lumborum Block vs. a TAP-block for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB3384
Record Dates: First submitted 2017-01-03; First posted 2017-01-18 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Inguinal Hernia; Pain, Postoperative
Keywords: Anterior Quadratus Lumborum block; Transversus Abdominis block; Truncal block
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Oxycodone; Ondansetron; Droperidol; Ropivacaine

STUDY DESIGN:
Intervention Model Description: * Group QLB: Anterior Quadratus Lumborum Block using ropivacaine 7,5 mg/ml, 20ml. Subcutaneous wound infiltration in all patients with ropivacaine 5 mg/ml,10 ml.
  * Group TAP: Transversus abdominis plane block using ropivacaine 7,5 mg/ml, 20 ml Subcutaneous wound infiltration in all patients with ropivacaine 5 mg/ml,10 ml.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Computer generated randomization with allocation in opaque envelopes. Randomization performed by other study personell than care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transmuscular Quadratus lumborum Block (Active Comparator): A single shot unilateral transmuscular Quadratus lumborum Block with Ropivacaine 7,5 mg/ml, 20 ml
  Interventions: Drug: Oksykodonhydroklorid; Drug: Ondansetron and Droperidol; Drug: Ropivacaine
- TAP Block (Active Comparator): A single shot unilateral TAP block with Ropivacaine 7,5 mg/ml, 20 ml
  Interventions: Drug: Oksykodonhydroklorid; Drug: Ondansetron and Droperidol; Drug: Ropivacaine

INTERVENTIONS:
Drug: Oksykodonhydroklorid — Oksykodonhydroklorid, 5 - 10 mg intravenously or orally postoperatively to reduce pain. Repetition until effect.
  Other Names: oxycodone
Drug: Ondansetron and Droperidol — When nausea and vomiting: Ondansetron 4mg and droperidol 0,625 mg intravenously
  Other Names: Ondansetron and Dridol
Drug: Ropivacaine — Local anesthetic for the block

SUMMARY:
One of the most common complications after hernia repair is postoperative and chronic pain. TAP (transverse abdominis plain) block is a recommended multimodal method of reducing postoperative pain in laparoscopic and open inguinal hernia repair. The objective of this study is to determine whether the use of a perioperative echo guided unilateral TAP block has a superior effect on postoperative pain after laparoscopic inguinal repair compared to an anterior Quadratus Lumborum Block with a long acting local anesthetic.

DETAILED DESCRIPTION:
One of the most common complications after hernia repair is postoperative and chronic pain. Postoperative pain is an expected but undesirable effect after an operation, which can result in an prolonged hospital stay or longer time to return fully to normal daily activities. There are indications that an insufficient treatment of postoperative pain is a risk factor for persistent or chronic pain after open and laparoscopic inguinal hernia repair (Berndsen FH 2007) (Nienhuijs SW 2005).

TAP (transverse abdominis plain) block is a recommended multimodal method of reducing postoperative pain in laparoscopic and open surgery (El-Dawlatly AA 2009; 102). TAP block (Meyer A 2015) and an anterior Quadratus Lumborum Block (Adhikary, S.D. 2017) are both recommended for inguinal hernia repair. The objective of this study is to determine, whether the use of a perioperative echo guided unilateral TAP block has a superior effect on postoperative pain after laparoscopic inguinal repair compared to the anterior Quadratus Lumborum Block with a long acting local anesthetic. There will be no further analysis in this study regarding the evidence of open hernia inguinal repair and chronic pain.

The primary endpoint:

Opioid consumption measured in orale morphine equivalents four hours postoperative.

The secondary endpoints:

Opoioid consumption measured in orale morphine equivalents after 24 hours, 48 hours and seven days postoperative.

Postoperative nausea and vomiting measured on a NRS scale 0-3 at timepoints 1,2,3 hours, 24 hours, 48 hours and 7 days. Sedation scores measured on a NRS scale 0-3 at timepoints 1,2,3 hours, 24 hours, 48 hours and 7 days. .

There will be conducted a telephone interview by a blinded study nurse at 24 h, 48 h and 7 days, interviewing the patients as to their NRS score, nausea, sedation, level of activity and satisfaction with their overall treatment.

Power and Sample Size Calculator A pilot consisting of 12 patients was performed. The patients recieved a TAP block before a elective laparoscopic inguinal hernia repair. The mean oral morphine equivalents after four hours postoperative was 8.75 mg and the standard deviation 5.93 mg. With a significant clinical difference of 50%,an α = 0,05 and an effect size of 80% (β = 0,2) the total sample size is 60 patients with 30 patients in each group.

Premedication: Paracetamol by weight (2 grams (g)>70 kilos (kg) <70 years, 1,5 g <70 kg >70 years, 1 g <50 kg) , Diclofenac by weight (100 milligrams (mg) >70 kg <70 years, 50 mg <70 kg >70 years).

General anaesthesia: TCI (Target Control Infusion = Anesthesia protocol): Propofol and Remifentanil Surgical procedure: Laparoscopic inguinal hernia repair. 5 mg/ml 10 ml Ropivacaine in the ports peroperatively.

Postoperatively:

* Oral paracetamol 1000 mg every 6 h
* In case of insufficient analgesia (NRS≥4) oxycodon 2-5 mg will be administered by a postoperative nurse.
* When nausea and vomiting occurs postoperatively, ondansetron 4 mg IV administers as the drug of first choice followed by droperidol 0,625 mg IV if the nausea/vomiting persists.

ELIGIBILITY:
Inclusion criteria;

* Age > 18 years
* BMI (body mass index) 20-35
* ASA (American Association of Anesthesiologists Classification system for physical status) I-III.
* Scheduled for elective laparoscopic inguinal hernia operation

Exclusion criteria:

* Allergy to latex, local anesthesia or opioids
* Chronic pain with daily opiate use
* Patients with severe renal and/or hepatic disease
* Local infection at the site of injection
* Systemic infection
* AV block 2-3
* Inability to understand written or spoken Norwegian
* Inability to cooperate
* Dementia
* Known abuse of alcohol or medication
* Coagulation disorder
* Pregnancy Previously operated with same side operation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption measured as orale morphine equivalents. | 0 - 4 hours
  Differences in opioid consumption after four hours.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 0 - 7 days postoperative.
  Nausea is measured by a NRS score 0-3 at the timepoints 1,2,3 hours, 24 hours, 48 hours and 7 days.
Sedation scores | 0 - 7 days postoperative.
  Sedation is measured by a NRS score 0-3 at the timepoints 1,2,3 hours, 24 hours, 48 hours and 7 days.
Opioid consumption measured in orale morphine equivalents. | 4 hours- 7 days postopertive.
  Opioid consumption measured at 24 hours, 48 hours and seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sverre Vamnes, MD, Ph.D., Study Chair — Senior consultant
Locations (1):
- Ostfold Hospital Trust, Moss, Moss, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Undecided
No sharing plan so far

REFERENCES:
- [Background] Berndsen FH, Petersson U, Arvidsson D, Leijonmarck CE, Rudberg C, Smedberg S, Montgomery A; SMIL Study Group. Discomfort five years after laparoscopic and Shouldice inguinal hernia repair: a randomised trial with 867 patients. A report from the SMIL study group. Hernia. 2007 Aug;11(4):307-13. doi: 10.1007/s10029-007-0214-7. Epub 2007 Apr 18. PMID 17440795
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Background] Meyer A, Bonnet L, Bourbon M, Blanc P. Totally extraperitoneal (TEP) endoscopic inguinal hernia repair with TAP (transversus abdominis plane) block as a day-case: a prospective cohort study. J Visc Surg. 2015 Jun;152(3):155-9. doi: 10.1016/j.jviscsurg.2014.12.005. Epub 2015 Jan 6. PMID 25575582
- [Background] Nienhuijs SW, Boelens OB, Strobbe LJ. Pain after anterior mesh hernia repair. J Am Coll Surg. 2005 Jun;200(6):885-9. doi: 10.1016/j.jamcollsurg.2005.02.005. PMID 15922201
- [Background] Petersen PL, Mathiesen O, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB. The effect of transversus abdominis plane block or local anaesthetic infiltration in inguinal hernia repair: a randomised clinical trial. Eur J Anaesthesiol. 2013 Jul;30(7):415-21. doi: 10.1097/EJA.0b013e32835fc86f. PMID 23549122
- [Background] Adhikary SD, El-Boghdadly K, Nasralah Z, Sarwani N, Nixon AM, Chin KJ. A radiologic and anatomic assessment of injectate spread following transmuscular quadratus lumborum block in cadavers. Anaesthesia. 2017 Jan;72(1):73-79. doi: 10.1111/anae.13647. Epub 2016 Oct 12. PMID 27730633